CLINICAL TRIAL: NCT06879262
Title: Clinical Study of Novel TLR2-Containing CAR-T Cells Targeting CD19 and CD22 for Refractory/Relapsed B-Cell Acute Lymphoblastic Leukemia and Non-Hodgkin Lymphoma
Brief Title: Clinical Study of Novel TLR2-Containing CAR-T Cells Targeting CD19 and CD22 for Relapsed/Refractory B-ALL and NHL
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Jia Wei, professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB202502060
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: R/R NHL
Keywords: CAR-T; CAR1922T2 T cells
MeSH Terms: interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Administer a single infusion of CAR1922T2 T cells to this group of patients following fludarabine plus cyclophosphamide (F+C) lymphodepletion, and conduct follow-up surveys at the required time points within three years post-infusion according to the visit schedule.
  Interventions: Biological: CAR1922T2 T cells（Targeting CD19 and CD22 with CAR-T cells）

INTERVENTIONS:
Biological: CAR1922T2 T cells（Targeting CD19 and CD22 with CAR-T cells） — Administer a single infusion of CAR1922T2 T cells to this group of patients following fludarabine plus cyclophosphamide (F+C) lymphodepletion

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and efficacy of CAR1922T2 T-cell therapy in participants with relapsed/refractory B-cell acute lymphoblastic leukemia and non-Hodgkin's lymphoma. Participants will receive a single infusion of CAR1922T2 T-cells and complete follow-ups over the next three years.

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia (ALL) is a hematological malignancy characterized by the clonal proliferation of precursor lymphoid cells, with a cure rate of only 30-40% in adults through standardized chemotherapy. Non-Hodgkin's lymphoma (NHL) is a highly heterogeneous group of lymphatic and reticular neoplasms derived from the clonal malignant proliferation of lymphoid cells, with 30-40% of patients developing into refractory disease or relapsing after initial treatment. Although CAR-T cell therapy targeting CD19 has made significant progress in the treatment of patients with refractory/relapsed B-cell acute lymphoblastic leukemia and non-Hodgkin's lymphoma, more than 50% of patients treated with CAR19 experience disease progression, which is related to the loss of CD19 on the cell surface. Therefore, our research team has developed a dual-specific CAR-T cell targeting both CD19 and CD22 to enhance the tumor-killing ability of CAR-T cells.

This clinical trial aims to evaluate the effectiveness and safety of CAR-T cell therapy targeting CD19 and CD22 (CAR1922T2 T cells) in participants with refractory/relapsed B-cell acute lymphoblastic leukemia and non-Hodgkin's lymphoma. After treatment with CAR1922T2 T cells, the effectiveness and safety of CAR1922T2 T-cell therapy for refractory/relapsed B-cell acute lymphoblastic leukemia and non-Hodgkin's lymphoma will be assessed through clinical symptom evaluation, quality of life assessment, biomarker testing, laboratory testing, imaging evaluation, adverse event monitoring, and follow-up surveys.

ELIGIBILITY:
Inclusion Criteria:

* 1. The patient or their legal guardian voluntarily participates and signs an informed consent form.

  2.Age between 18-80 years old (inclusive), with no gender restrictions. 3.Diagnosed with acute B-cell acute lymphoblastic leukemia or non-Hodgkin's lymphoma according to the WHO 2016 classification.

  4.CD19 or CD22 positivity confirmed by flow cytometry or histopathology. 5.Diagnosed with refractory/relapsed B-cell acute lymphoblastic leukemia or non-Hodgkin's lymphoma.

  6.Good major organ function:
  1. Liver function: ALT/AST < 3 times the upper limit of normal (ULN) and total bilirubin ≤ 34.2 μmol/L;
  2. Kidney function: Creatinine clearance rate (Cockcroft-Gault method) ≥ 60 mL/min;
  3. Lung function: Oxygen saturation ≥ 95%, with no active pulmonary infection;
  4. Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%; no significant pericardial effusion, no clinically significant ECG abnormalities.

     7.Women of childbearing age with negative urine/blood pregnancy test during screening and agree to use contraceptive measures for at least 1 year after infusion; male subjects with reproductive capacity must agree to use effective barrier contraceptive methods for at least 1 year after infusion.

     8.ECOG score ≤ 1. 9.Life expectancy greater than 3 months.

     Exclusion Criteria:
* 1.Women who are breastfeeding. 2.Patients with uncontrollable infectious diseases within 4 weeks before enrollment.

  3.Active hepatitis B/C. 4.HIV-infected patients. 5.Patients with severe autoimmune diseases or immunodeficiency diseases. 6.Patients with allergic constitution, allergic to antibodies or cytokines and other large molecule biological drugs.

  7.Patients who have participated in other clinical trials within 4 weeks before enrollment.

  8.History of clinically significant central nervous system diseases: such as epilepsy, paralysis, aphasia, stroke, severe brain trauma, dementia, Parkinson's disease, cerebellar diseases, organic brain syndromes.

  9.Patients with mental illness. 10.Patients with drug abuse/addiction. 11.Use of contraindicated medications.
  1. . Steroids: Use of therapeutic doses of corticosteroids (defined as prednisone or equivalent >20 mg/day) within 7 days before leukocyte collection, or within 72 hours before CAR-T cell infusion targeting CD19 and CD22. However, physiological replacement, topical, and inhaled corticosteroids are allowed.
  2. . Chemotherapy: Received salvage chemotherapy within 2 weeks before leukocyte collection.
  3. . Allogeneic cell therapy: Received donor lymphocyte infusion within 4 weeks before leukocyte collection.
  4. . GVHD treatment: Received anti-GVHD treatment within 4 weeks before CAR-T cell infusion targeting CD19 and CD22.
  5. . Use of alemtuzumab, or cladribine within 6 months before leukocyte collection, or use of chlorambucil or clofarabine within 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
ORR | 3 years
  The overall response rate (ORR) includes both complete response (CR) and partial response (PR), and uses the Clopper-Pearson method to calculate the two-sided 95% confidence interval.

IPD SHARING:
Plan to Share IPD: No